CLINICAL TRIAL: NCT03748589
Title: Application of I-gel Laryngeal Mask Airway in Infants and Children Undergoing Surgical Procedures
Brief Title: Application of I-gel Laryngeal Mask Airway in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xian Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018008
Record Dates: First submitted 2018-10-24; First posted 2018-11-21 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2018-12

CONDITIONS: the Efficacy and Performance of the Pediatric I-gel Mask
Keywords: i-gel; pediatric; laryngeal mask airway; children
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- airway type 1 (Experimental): The children weighed between 2-5kg are assigned into this group,they are allocated with i-gel laryngeal mask airway type 1
  Interventions: Device: laryngeal mask airway
- airway type 1.5 (Experimental): The children weighed between 5-12kg are assigned into this group,they are allocated with i-gel laryngeal mask airway type 1.5
  Interventions: Device: laryngeal mask airway
- airway type 2 (Experimental): The children weighed between 10-25kg are assigned into this group,they are allocated with i-gel laryngeal mask airway type 2
  Interventions: Device: laryngeal mask airway
- airway type 2.5 (Experimental): The children weighed between 25-35kg are assigned into this group,they are allocated with i-gel laryngeal mask airway type 2.5
  Interventions: Device: laryngeal mask airway

INTERVENTIONS:
Device: laryngeal mask airway — i-gel laryngeal mask airway is a supraglottic airway device made from a medical grade thermoplastic elastomer , is a non-inflatable device to create anatomical seal of the pharyngeal, laryngeal and perilaryngeal structures and avoid compression trauma.
  Other Names: i-gel

SUMMARY:
Background The laryngeal mask airway (LMA) is a supraglottic airway device ,which is commonly used to manage children's airways, because it is typically easy to use and can avoid problems specific to tracheal intubation. Since the LMA was introduced into clinical practice in 1988 , various types of LMAs have been developed, the safety and efficacy of which have been established in both adults and children.The paediatric i-gel is a relatively new and disposable supraglottic airway device for children, which is made of a soft gel-like elastomer with a non-inflatable cuff and a channel for gastric catheter placement . It does not require cuff inflation ,reducing the complications associated with compression trauma and high cuff pressure . Medical-grade thermoplastic elastomer creates a more intimate interface for interacting with supraglottic tissue. The usage of i-gel mask is more common in adults ,though a large scale study focusing on children is lacking.

Objectives:

To evaluate the efficacy and performance of the pediatric i-gel mask

Methods:

From November 2018 to March 2019, subjects are selected from patients who undergo elective surgery at Xi'an Children's Hospital, within the age of 0 to 108 months old, with an American Society of Anesthesiologists physical status I or II .They were assigned into four groups according to their weight. Four groups are : 2-5 kg (group 1#), 5.1-12.0 kg (group 1.5#), 10-25kg (group 2#) 25-35kg(group 2.5#). The primary outcome is the clinical performance of the airways: the rate of insertion at first attempt,the ease of insertion,the insertion time,the oropharyngeal leak pressure(OLP),the fibreoptic view and the ease of gastric tube insertion. The secondary outcome is the frequency of other perioperative complications as listed in the detail information section.

DETAILED DESCRIPTION:
methods This is a prospective, randomized, parallel-group, single sample study ,which was approved by the Ethics Committee of Children's Hospital affiliated to Xi'an Jiaotong University.The experiment is expected to be completed between December 2018 and March 2019 in Xi'an children's Hospital, signed consent will be obtained from the parents or the guardian of the child participating in the study.The inclusion criteria are: children aged between 0 to 108 months, Weighed between 2 to 35 kg,with an American Standards Association (ASA )physical status Ι or Ⅱ, who are scheduled for elective surgery shorter than four hours under general anesthesia . In addition,the operation of supraglottic airway devices needs to be seamless during perioperative period. Children with below condition will be excluded form the experiment:a suspected difficult airway, a history of upper respiratory tract infection two weeks before operation ,being at risk of aspiration (such as non-fasting status , gastroesophageal reflux disease and hiatus hernia),lung diseases, limited head-neck movements, and those refusing to participate.The children with symptoms bradycardia and conduction block shown on EEG are also excluded from this experiment.The children were assigned into four groups based on their weights : size 1 for 2-5kg ,size 1.5 for 5-12 kg, size 2 for 10-25 kg, size 2.5 for 25-35 kg . The required device is prepared according to the child's weight and using the the manufacturer's guidelines . The children's group allocation were operated by a researcher who do not participate in post anesthesia care unit or outcome assessment. All children involved in the experiment, the children's parents, and the data analyzer are blind to the device used. In preparation for surgery,children are fasted 8h from solid food with fat content, 6h from semi-solid food and liquid food ,4h for breast milk and 2 h for clear water .Premedication is provided about 20 minutes before entering the operating room, by which children receive intranasal dexmedetomidine 1.5ug/kg, so that children can enter the operating room quietly. On arrival in the operating room, children were monitored using pulse oximetry, electrocardiography, non-invasive blood pressure, and capnography. General anaesthesia was induced with 100% oxygen 2-4 Liter(L)/min. Injection atropine 0.01mg/kg、fentanyl 2 μg/kg 、 propofol 2mg/kg 、vecuronium bromide 0.1 mg/kg intravenously (IV) in turn.After loss of consciousness, children are promptly positioned supine with an adequate sized roll underneath the neck to establish optimal position.Achieving appropriate anesthesia depth,children are randomised to have inserted i-gel ,The jaw thrust maneuver are used to confirm anesthesia depth whether it is suitable for placing the laryngeal mask and facilitating its placement. We do not administer neuromuscular blocking during intraoperative period. Two anesthesiologists came to the hospital for working at least one year and experienced in inserting supraglottic airway devices in at least 200 pediatric patients. The device was inserted according to the manufacturer's recommendations .Device insertion was considered successful by observing bilateral chest wall movement,as well as a stable square-wave capnogram trace ,the lung breath sound with no audible leak .Three failed insertion attempts are considered failed insertion of the device, and patients were withdrawn from the study.Tracheal intubation was considered after failure of three times of laryngeal mask airway placement.

Insertion time was measured from the moment a device was picked up until confirmation of the first wave on a capnogram，The ease of device placement was assessed using a subjective grading score of 1-4 (1: no resistance, 2: mild resistance, 3: moderate resistance, 4: inability to place the device) by the anesthesiologist. We also record the manipulations for improving device position, such as adjusting the insertion depth, conducting a jaw thrust maneuver, or flexion/extension of the head.

Oropharyngeal leak pressure and fiberoptic view through the device were assessed. Oropharyngeal leak pressure was determined by closing the adjustable pressure-limiting valve to 30 centimeter water column(cmH 2 O) at the fresh gas flow rate of 3 L/min, switching the mechanical ventilation to manual ventilation, and reading the airway pressure on the monitor in the anesthesia machine which an audible leak on auscultation over neck was defined as OLP. The OLP was not allowed to exceed 30 cmH 2 O to avoid barotrauma, If mean airway pressure is higher than OLP or insufficient ventilation (lesser than 5 ml/kg) occurred during the airway maintenance, proper manipulations (pushing or pulling of device, extension or flexion of the head, jaw thrust) were performed. If appropriate manipulation does not solve the problem, the device should be removed and endotracheal intubation be performed. The anatomical position of the LMA in relation to the glottis was evaluated by placing a fiberoptic bronchoscope through the device .The fiberoptic view is classified into four grades by observing the fiberoptic views (grade 1: vocal cords not visible, grade 2: vocal cords and anterior epiglottis visible, grade 3: vocal cords and posterior epiglottis visible, grade 4: only vocal cords visible). The 8-12 French size gastric tubes are used for those groups. A well-lubricated gastric tube is prepared before inserted into the stomach through gastric port of airway device. The assessment of correct placement is through detection of injected air by epigastric auscultation or by aspiration of gastric content .A grading scale(1:easy,2:difficult,3：failure) is used for assessing the ease of gastric tube insertion.Easy is defined as placing the tube successfully in the first attempt,difficult is defined as placing the tube successfully within two attempts, failure is defined as inability to establish correct placement within three placements.Anesthesia was maintained using 2%~3% sevoflurane and remifentanil 0.2~0.4ug/kg•min.1 ug/kg fentanyl is added again before the skin incision and suture. At the end of surgery, the anesthetics are terminated. The patient was then moved to the postanesthesia care unit (PACU).We recorded heart rate, mean blood pressure, oxygen saturation, peak inspiratory pressure and complications during the induction and maintenance of anesthesia. At the conclusion of the surgery, when the tidal volume is >6 ml/kg or end-tidal carbon dioxide(CO2) is less than 50 mmHg,we can stop the mechanical ventilation and keep the patient's spontaneous respiration. The LMA is removed when evidence of adequate emergence including spontaneous eye opening, grimacing using forehead and/or eyebrow, and purposeful movement. In addition,we also observed the complication such as coughing, bronchospasm, laryngospasm, desaturation (SpO 2 < 90%), regurgitation, aspiration, sore throat, blood-on LMA, postoperative nausea and vomiting (PONV), breath-holding and teeth or lip injury during anesthesia maintenance and emergence . A blinded investigator assessed all patients in the PACU and conducted a ward visit or telephone interview 24 h after the end of surgery. In our study, the primary outcome is oropharyngeal leak pressure，the secondary outcome are the rate of successful insertion at first attempt, fiberoptic view，insertion time，ease of insertion，ease of gastric tube insertion。 We recorded complications including coughing, breath-holding, desaturation, laryngospasm or bronchospasm，blood-on LMA, sore throat, postoperative nausea and vomiting (PONV), regurgitation, aspiration, teeth or lip injury.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 2 to 35 kg ASA physical status Ι or Ⅱ elective surgery operation time not longer than four hours general anesthesia

Exclusion Criteria:

* a history of upper respiratory tract infection two weeks before operation risk of aspiration (such as non-fasting status , gastroesophageal reflux disease and hiatus hernia) lung diseases limited head-neck movements those refusing to participate children whose EEG showing bradycardia and conduction block

Ages: 1 Day to 108 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 413 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | At 5 min after the insertion of i-gel protector
  reading the airway pressure on the monitor in the anesthesia machine

SECONDARY OUTCOMES:
insertion time | During the insertion of i-gel protector
  insertion time is measured from the moment of picking up the device to confirming the first the appearance of the ETCO2 on monitor screen
ease of insertion | during the insertion of i-gel protector
  Ease of insertion we are using a subjective grading score of 1-4 (1: requiring no additional maneuver, 2:requiring 1 additional maneuver, 3:requiring 2 additional maneuver, 4: requiring more than 3 maneuver)
fiberoptic view | At 15 min after the insertion of i-gel protector
  After insertion of the device, observe the accuracy of insertion location by the fiberoptic views through the device(grade 1: vocal cords not visible, grade 2: vocal cords and anterior epiglottis visible, grade 3: vocal cords and posterior epiglottis visible, grade 4: only vocal cords visible)
the rate of successful insertion at first attempt | During the first attempt insertion of i-gel protector
  the insertion is successful at first attempt
the ease of gastric tube insertion | At 25 min after the insertion of i-gel protector
  subjective grading scale(1:easy，2:difficult,3:failed insertion) is used for assessing the ease of gastric tube insertion.Easy is defined as placing the tube successfully in the first attempt,difficult is defined as placing the tube successfully within two attempts, failure is defined as inability to establish correct placement within three placements.

CONTACTS AND LOCATIONS:
Overall Officials: fang li yang, doctor, Study Chair — Xian Children's Hospital
Locations (1):
- Xi'an Children's Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banerjee G, Jain D, Bala I, Gandhi K, Samujh R. Comparison of the ProSeal laryngeal mask airway with the I-Gel in the different head-and-neck positions in anaesthetised paralysed children: A randomised controlled trial. Indian J Anaesth. 2018 Feb;62(2):103-108. doi: 10.4103/ija.IJA_594_17. PMID 29491514
- [Background] Lee YC, Yoon KS, Park SY, Choi SR, Chung CJ. A comparison of i-gel and Laryngeal Mask Airway Supreme during general anesthesia in infants. Korean J Anesthesiol. 2018 Feb;71(1):37-42. doi: 10.4097/kjae.2018.71.1.37. Epub 2017 Aug 14. PMID 29441173
- [Background] Alzahem AM, Aqil M, Alzahrani TA, Aljazaeri AH. Erratum: Ambu AuraOnce versus i-gel laryngeal mask airway in infants and children undergoing surgical procedures. A randomized controlled trial. Saudi Med J. 2017 Dec;38(12):1267. No abstract available. PMID 29209682
- [Background] Yang GZ, Xue FS, Li HX, Liu YY. Comparing i-gel and Ambu AuraOnce laryngeal mask airway in pediatric patients. Saudi Med J. 2017 Dec;38(12):1262-1263. doi: 10.15537/smj.2017.12.20856. PMID 29209679
- [Background] Bhattacharjee S, Som A, Maitra S. Comparison of LMA Supreme with i-gel and LMA ProSeal in children for airway management during general anaesthesia: A meta-analysis of randomized controlled trials. J Clin Anesth. 2017 Sep;41:5-10. doi: 10.1016/j.jclinane.2017.04.019. Epub 2017 Jun 1. PMID 28802606
- [Background] Park JH, Kim JY, Park K, Kil HK. A randomized comparison of volume- and pressure-controlled ventilation in children with the i-gel: Effects on peak inspiratory pressure, oropharyngeal leak pressure, and gastric insufflation. Medicine (Baltimore). 2017 May;96(18):e6772. doi: 10.1097/MD.0000000000006772. PMID 28471973
- [Background] Alzahem AM, Aqil M, Alzahrani TA, Aljazaeri AH. Ambu AuraOnce versus i-gel laryngeal mask airway in infants and children undergoing surgical procedures. A randomized controlled trial. Saudi Med J. 2017 May;38(5):482-490. doi: 10.15537/smj.2017.5.17960. PMID 28439597
- [Background] Jain D, Ghai B, Gandhi K, Banerjee G, Bala I, Samujh R. Evaluation of I-Gel size 2 airway in different degrees of neck flexion in anesthetized children - a prospective, self-controlled trial. Paediatr Anaesth. 2016 Dec;26(12):1136-1141. doi: 10.1111/pan.13001. Epub 2016 Oct 25. PMID 27779349
- [Background] Nirupa R, Gombar S, Ahuja V, Sharma P. A randomised trial to compare i-gel and ProSeal laryngeal mask airway for airway management in paediatric patients. Indian J Anaesth. 2016 Oct;60(10):726-731. doi: 10.4103/0019-5049.191670. PMID 27761035
- [Background] Gu Z, Jin Q, Liu J, Chen L. Observation of ventilation effects of I-gel, Supreme and Ambu AuraOnce with respiratory dynamics monitoring in small children. J Clin Monit Comput. 2017 Oct;31(5):1035-1041. doi: 10.1007/s10877-016-9917-6. Epub 2016 Aug 4. PMID 27492428
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989